CLINICAL TRIAL: NCT01154413
Title: Implementation of a Diabetes Management Protocol as Compared to Conventional Management in a Heart Hospital's Non-Intensive Care Unit: Randomized Clinical Trial
Brief Title: Implementation of a Diabetes Management Protocol as Compared to Conventional Management in a Heart Hospital's Non-Intensive Care Unit: Randomized Clinical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Maria Antonieta Pereira de Moraes, Instituto de Cardiologia Fundação Universitária de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP3984/07
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive education of the doctor/nursing team on the protocol (Experimental)
  Interventions: Behavioral: Intensive education of the doctor/nursing team on the protocol
- Without intervention in the team (No Intervention)
  Interventions: Behavioral: Intensive education of the doctor/nursing team on the protocol

INTERVENTIONS:
Behavioral: Intensive education of the doctor/nursing team on the protocol

SUMMARY:
To asses the effectiveness of implementing a diabetes management protocol (early insulinization, avoiding use of SSI) in a hearth hospital's non-intensive care unit.

DETAILED DESCRIPTION:
Management of diabetes in patients admitted to non-intensive unit of a cardiology hospital in order to reduce the number of episodes of hypo-and hyperglycemia, improve glucose control and reducing the number of hospital days.

Eligibility criteria:

Patients with previous history of diabetes mellitus type 2, or are in use of oral antidiabetics or insulin or having fasting glucose or less 126 mg / dL or random blood glucose greater 200 mg / dL in both sexes, aged greater 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Previous history of diabetes mellitus type 2, or they were using oral anti-diabetic or insulin had a fasting glucose greater than or equal to 126 mg / dL or random blood glucose greater 200 mg / dL in both sexes, age greater than or equal 18 years

Exclusion Criteria:

* Patients with known presence of cancer, while using corticosteroids, immunosuppressants on hemodialysis, with cognitive and neurological sequelae, patients whose admission had shorter duration than 72 hours, when they came transferred from intensive care units in other protocols using insulin when no doctor would agree to join the protocol and those who do not agree to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2007-12; Primary Completion 2007-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Reduction in hypo/hyperglycemia episodes

SECONDARY OUTCOMES:
Lower mean glycemia, reduced time of stay in hospital

REFERENCES:
- [Derived] Moraes MA, Rodrigues J, Cremonesi M, Polanczyk C, Schaan BD. Management of diabetes by a healthcare team in a cardiology unit: a randomized controlled trial. Clinics (Sao Paulo). 2013 Nov;68(11):1400-7. doi: 10.6061/clinics/2013(11)03. PMID 24270950